CLINICAL TRIAL: NCT06037109
Title: VIDAS® NEPHROCLEAR CCL14 Reference Interval Study
Brief Title: VIDAS® NEPHROCLEAR Reference Interval Study
Status: Completed | Type: Observational
Sponsor: BioMérieux (Industry)
Responsible Party: Sponsor
Other Study IDs: B3166-CTPR03
Record Dates: First submitted 2023-09-07; First posted 2023-09-14 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2023-09

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Urine samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

GROUPS / COHORTS (2):
- Apparently Healthy Adults: Apparently healthy adults (age ≥ 21 years); who have provided written informed consent for sample use in this study
  Interventions: Device: Diagnostic Test: VIDAS® NEPHROCLEAR™ CCL14 Test
- Adults with Chronic, Stable Morbidities: Adults (age ≥ 21 years);with one or more of the following chronic, stable morbid conditions.
  Interventions: Device: Diagnostic Test: VIDAS® NEPHROCLEAR™ CCL14 Test

INTERVENTIONS:
Device: Diagnostic Test: VIDAS® NEPHROCLEAR™ CCL14 Test — Previously collected urine samples will be tested using the VIDAS® NEPHROCLEAR™ CCL14 Test

SUMMARY:
This is a multi-center sample analysis study in which urine samples previously collected from apparently healthy adult subjects, and subjects with stable chronic morbidities but without AKI in order to establish the reference range for the VIDAS® NEPHROCLEAR™ CCL14 test.

DETAILED DESCRIPTION:
The VIDAS® NEPHROCLEAR™ CCL14 Test is intended to be used in conjunction with clinical evaluation, in ICU patients with moderate to severe (stage 2 or 3) acute kidney injury (AKI), as an aid in the risk assessment for developing persistent severe AKI (stage 3 AKI lasting ≥ 72 hours) within 48 hours of patient assessment.

The VIDAS® NEPHROCLEAR™ CCL14 Test is intended to be used in patients 21 years of age or older.

The objective of this study is to determine the reference range for CCL14 concentration in Apparently Healthy Adults and Adults with Chronic, Stable Morbidities

ELIGIBILITY:
Cohort A

Inclusion Criteria:

* Apparently healthy adults (age ≥ 21 years);
* Provide written informed consent for study (AST-017) participation

Exclusion Criteria:

* Any known or suspected acute illness or condition - including acute infections - at the time of enrollment or within the previous 30 days;
* Any known or suspected significant new onset or chronic morbid medical condition such as:
* Active cancer
* Arrhythmia (atrial fibrillation, heart block, ventricular tachycardia)
* Chronic coagulation abnormality
* Chronic obstructive pulmonary disease (including emphysema, chronic bronchitis, and asthma)
* Chronic pancreatitis
* Chronic renal insufficiency
* Congestive heart failure
* Coronary artery disease
* Diabetes mellitus (Type 1 or Type 2)
* Gout
* Hyper- or hypothyroidism
* Hyperlipidemia (includes hypercholesterolemia)
* Hypertension
* Immunocompromised
* Inflammatory bowel disease (including Crohn's disease and ulcerative colitis)
* Liver cirrhosis
* Neuromuscular disease
* Peripheral vascular disease (a.k.a. peripheral artery disease)
* Polycystic kidney disease
* Rheumatoid arthritis
* Systemic Lupus Erythematosus
* Trauma-related surgery within the last 6 months;
* Any surgery, hospitalization or institutionalization (such as in a nursing home) during the previous 3 months;
* Received any blood product transfusion within the previous 2 months;
* Pregnant women or children;
* Prisoners or institutionalized individuals;
* Already provided a urine sample for the AST-017 study

Cohort B

Inclusion Criteria:

* Adults (age ≥ 21 years);
* One or more of the following chronic, stable morbid conditions:
* Active cancer
* Arrhythmia (atrial fibrillation, heart block, ventricular tachycardia)
* Chronic coagulation abnormality
* Chronic obstructive pulmonary disease (including emphysema, chronic bronchitis, and asthma)
* Chronic pancreatitis
* Chronic renal insufficiency
* Congestive heart failure
* Coronary artery disease
* Diabetes mellitus (Type 1 or Type 2)
* Gout
* Hyper- or hypothyroidism
* Hyperlipidemia (includes hypercholesterolemia)
* Hypertension
* Immunocompromised
* Inflammatory bowel disease (including Crohn's disease and ulcerative colitis)
* Liver cirrhosis
* Neuromuscular disease
* Peripheral vascular disease (a.k.a. peripheral artery disease)
* Polycystic kidney disease
* Rheumatoid arthritis
* Systemic Lupus Erythematosus
* Provide written informed consent for study participation.
* For Cohort B subjects in the AST-017 Study:
* Subjects were considered to have the above condition(s) if he/she had the diagnosis by a healthcare professional and/or was under treatment by a healthcare professional for the listed condition(s).
* Subjects with a condition (e.g., hypertension, hypercholesterolemia) controlled by medications were enrolled.
* To be considered chronic and stable, the condition(s) must have been present for at least 1 year and without any acute change (decompensation or improvement) within the 3 months prior to enrollment.

Exclusion Criteria:

* Any known or suspected acute illness or condition - including acute infections - at the time of enrollment or within the previous 30 days;
* Any new onset or unstable morbidities;
* Trauma-related surgery within the last 6 months;
* Any surgery, hospitalization or institutionalization (such as in a nursing home) during the previous 3 months;
* Received any blood product transfusion within the previous 2 months;
* Pregnant women or children;
* Prisoners or institutionalized individuals;
* Already provided a urine sample for this (AST-017) study.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Samples were collected from apparently healthy adults (n = ~300) and adults with pre-specified underlying chronic stable morbidities (n = ~300).
Sampling Method: Non-Probability Sample
Enrollment: 585 (Actual)
Dates: Start 2023-07-18 (Actual); Primary Completion 2023-12-28 (Actual); Study Completion 2023-12-28 (Actual)

PRIMARY OUTCOMES:
CCL14 concentration in urine | Samples tested within 2 years of collection
  CCL14 concentration will be measured using the VIDAS Necphroclear CCL14 Assay

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - George Washington University, Washington D.C., District of Columbia
  - University of Illinois Chicago, Chicago, Illinois

IPD SHARING:
Plan to Share IPD: No